CLINICAL TRIAL: NCT02801331
Title: A Randomized Controlled Study of Stochastic Vibrotactile Stimulation for Neonatal Abstinence Syndrome: Therapeutic Efficacy and Neurobehavioral Outcomes
Brief Title: Efficacy and Outcomes of a Non-Pharmacological Intervention for Neonatal Abstinence Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elisabeth B Salisbury (Other)
Collaborators: University of Pittsburgh (Other); National Institute on Drug Abuse (NIDA) (NIH); University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor-Investigator, Elisabeth B Salisbury, Visiting Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY21040054; 1R01DA042074-01 (NIH)
Record Dates: First submitted 2016-06-09; First posted 2016-06-15 (Estimated); Results first posted 2024-05-23 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: Stochastic Resonance; Fetus/Newborn Infant; Drug Withdrawal; Substance Abuse
MeSH Terms: conditions — Neonatal Abstinence Syndrome; Substance Withdrawal Syndrome; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Stochastic Vibrotactile Stimulation (SVS) (Experimental): Infants randomized to this arm will receive daily intervals of continuous SVS (ON) and no SVS (OFF) throughout hospitalization, starting within 48-hrs post birth. SVS will be complementary to standard of clinical care (e.g., clinically-determined pharmacological management; routine parental/volunteer holding; breast and/or bottle feed).
  Interventions: Device: Stochastic Vibrotactile Stimulation (SVS)
- Treatment as Usual (TAU) (No Intervention): Infants randomized to this arm will be enrolled within 48-hours post birth and receive treatment as usual (TAU)- standard of clinical care (e.g., clinically-determined pharmacological management, routine/volunteer holding; breast and/or bottle feed). Infants will not receive any SVS.

INTERVENTIONS:
Device: Stochastic Vibrotactile Stimulation (SVS) — Infant crib mattress will be replaced with a specially constructed mattress (non-commercially available) to provide gentle, stochastic vibration during mattress stimulations.
  Arms: Stochastic Vibrotactile Stimulation (SVS)

SUMMARY:
The purpose of this study is to examine the efficacy of a specially-constructed crib mattress that delivers gentle vibrations (stochastic vibrotactile stimulation) as a complementary, non-pharmacological intervention for treating drug withdrawal in newborns exposed to opioids in utero.

DETAILED DESCRIPTION:
This study will test the therapeutic efficacy of stochastic vibrotactile stimulation (SVS) for reducing withdrawal symptoms, pharmacological treatment and hospitalization, and for improving neurobehavioral developmental outcomes in opioid-exposed newborns.

Candidates at-risk for NAS due opioid exposure in utero will be identified to investigators by medical caregiver and/or prescreened using HIPAA Waiver for recruitment (maternal-prenatal; infant-postnatal). Infants will be randomized into either SVS (complementary to standard of care) or Treatment as Usual (TAU), restricted by equipment (mattress) availability. Infants will be enrolled and assigned to a condition within 48 hours post birth and participate throughout hospitalization. Infants assigned SVS will receive daily intervention of continuous intervals of SVS throughout hospitalization using a specially constructed crib mattress that delivers gentle vibrations at preset intervals.

Specific Aim 1. Determine the efficacy of SVS as a non-pharmacological therapy complementary to standard of care for reducing severity and duration of opioid withdrawal in newborns compared to TAU alone. Quantify clinical variables: NAS severity, treatment days, days in hospital, velocity of weight gain, cumulative morphine dose.

Specific Aim 2. Compare neurobehavioral outcomes in fetal drug-exposed infants between infants who received SVS and those who received TAU. Longitudinal outcomes assessment at 6-months and 1 year to test whether early intervention with SVS compared to standard care improves physical, social, emotional and cognitive development.

ELIGIBILITY:
Inclusion Criteria: Eligible subjects are infants currently in the NICU or Newborn Nursery at University of Massachusetts Memorial Hospital or at Magee Women's Hospital of UPMC and:

* Full-term infants (≥37 wks gestational age)
* Newborns at risk for NAS due to opioid-exposure in utero
* At-risk infants will be infants who present with confirmed meconium and/or urine toxicology report and/or documented medical record for opioids (e.g., methadone, buprenorphine/subutex, oxycodone, heroin); may also have prenatal exposure to benzodiazepines, barbiturates, amphetamines, cannabinoids, alcohol, nicotine and/or caffeine.

Exclusion Criteria: Eligible infants meeting the inclusion criteria above will be excluded from participation in the study if he/she:

* Born less than <37weeks.
* Has a clinically significant congenital abnormality
* Has a clinically significant fetal anomaly
* Has hydrocephalus or intraventricular hemorrhage >grade 2
* Has a seizure disorder not related to drug withdrawal
* Has a clinically significant cardiac shunt
* Has anemia (hemoglobin<8g/dL)
* Requires mechanical respiratory support
* Has MRSA or infection at time of the study

Ages: 1 Hour to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 208 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth B Salisbury, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bloch-Salisbury E, Bogen D, Vining M, Netherton D, Rodriguez N, Bruch T, Burns C, Erceg E, Glidden B, Ayturk D, Aurora S, Yanowitz T, Barton B, Beers S. Study design and rationale for a randomized controlled trial to assess effectiveness of stochastic vibrotactile mattress stimulation versus standard non-oscillating crib mattress for treating hospitalized opioid-exposed newborns. Contemp Clin Trials Commun. 2021 Feb 11;21:100737. doi: 10.1016/j.conctc.2021.100737. eCollection 2021 Mar. PMID 33748529
- [Background] Bloch-Salisbury E, Rodriguez N, Bruch T, McKenna L, Goldschmidt L. Physiologic dysregulation in newborns with prenatal opioid exposure: Cardiac, respiratory and movement activity. Neurotoxicol Teratol. 2022 Jul-Aug;92:107105. doi: 10.1016/j.ntt.2022.107105. Epub 2022 May 27. PMID 35636580
- [Background] Liu VY, Flahive JM, Bloch-Salisbury E. Actigraphy: An Adjunctive Method to Measure Irritability in Opioid-Exposed Newborns. J Nurs Meas. 2024 Oct 24;32(3):467-476. doi: 10.1891/JNM-2023-0020. PMID 37353324
- [Result] Bloch-Salisbury E, Wilson JD, Rodriguez N, Bruch T, McKenna L, Derbin M, Glidden B, Ayturk D, Aurora S, Yanowitz T, Barton B, Vining M, Beers SR, Bogen DL. Efficacy of a Vibrating Crib Mattress to Reduce Pharmacologic Treatment in Opioid-Exposed Newborns: A Randomized Clinical Trial. JAMA Pediatr. 2023 Jul 1;177(7):665-674. doi: 10.1001/jamapediatrics.2023.1077. PMID 37184872
- [Derived] Pahl A, Young L, Buus-Frank ME, Marcellus L, Soll R. Non-pharmacological care for opioid withdrawal in newborns. Cochrane Database Syst Rev. 2020 Dec 21;12(12):CD013217. doi: 10.1002/14651858.CD013217.pub2. PMID 33348423
- See also: Study design and rationale for a randomized controlled trial to assess effectiveness... — https://pubmed.ncbi.nlm.nih.gov/33748529/
- See also: Physiologic dysregulation in newborns with prenatal opioid exposure: Cardiac, respiratory and movement activity — https://pubmed.ncbi.nlm.nih.gov/35636580/
- See also: Actigraphy: An Adjunctive Method to Measure Irritability in Opioid-Exposed Newborns — https://pubmed.ncbi.nlm.nih.gov/37353324/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants recruited at UMass between March 9, 2017 and February 25, 2020; Infants recruited at Pitt between and August 18, 2017 and March 10, 2020.
  Enrollment was terminated early due to Covid-19 in-person study restrictions and unanticipated reduction and relocation of project personnel (208 recruited/220 anticipated enrollment).
Period: Overall Study
Arm/Group | Stochastic Vibrotactile Stimulation (SVS) | Treatment as Usual (TAU)
Started (mITT-reflects treatment received) | 105 | 103
Completed (Completed hospitalization at respective site (does not include post-hospitalization followup)) | 94 | 87
Not Completed | 11 | 16
Not completed — Transferred to another hospital | 8 | 7
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Subsequently met exclusion/withdrawal criteria | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stochastic Vibrotactile Stimulation (SVS) | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 105 | 103 | 208
Age, Continuous [Mean (Standard Deviation); unit: weeks] — gestational age (weeks)
  weeks | 39.1 (1.2) | 38.9 (1.2) | 39.0 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 57 | 115
  Male | 47 | 46 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 11 | 21
  Not Hispanic or Latino | 90 | 85 | 175
  Unknown or Not Reported | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 2 | 6
  White | 75 | 78 | 153
  More than one race | 19 | 17 | 36
  Unknown or Not Reported | 6 | 6 | 12
Birthweight [Mean (Standard Deviation); unit: grams] | 3081 (528) | 3054 (445) | 3068 (488)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Administered Morphine Treatment
Description: Number of infants treated with morphine (first line pharmacotherapy at both sites).
  Number of infants who received pharmacotherapy (met clinical criteria to treat), index of NAS severity (per Finnegan scores).
Time Frame: Participants will be monitored for the duration of their newborn nursery stay, which is an expected mean of 7 days
Population: Analyzed infants: completed hospitalization at respective study site
Measure: Count of Participants; unit: Participants
Arm/Group | Stochastic Vibrotactile Stimulation (SVS) | Treatment as Usual (TAU)
Number analyzed (Participants) | 94 | 87
Participants | 29 | 31
Statistical Analysis 1: Comparison: Stochastic Vibrotactile Stimulation (SVS) vs Treatment as Usual (TAU); Test type: Equivalence — A test of equivalence was conducted for unadjusted comparisons. A chi squared test of proportions was used for unadjusted comparisons; p = .60, Chi-squared — Unadjusted

2. Primary Outcome: Cumulative Pharmacological Treatment- Morphine Dose
Description: Normalized cumulative morphine dose for infants who completed treatment at respective hospital site (mg/kg).
Time Frame: Participants will be monitored for the duration of their hospitalization, which is an expected mean of 21 days
Population: Analyzed cohort who received morphine treatment
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Stochastic Vibrotactile Stimulation (SVS) | Treatment as Usual (TAU)
Number analyzed (Participants) | 29 | 31
mg/kg | 7.3 (6.6) | 8.2 (7.5)
Statistical Analysis 1: Comparison: Stochastic Vibrotactile Stimulation (SVS) vs Treatment as Usual (TAU); Test type: Equivalence — A statistical test comparing cumulative morphine dose was performed for the cohort that was treated with morphine (n=60); p = .62, t-test, 2 sided; degrees of freedom =58 for cohort analyzed that received morphine treatment

3. Primary Outcome: Hospitalization Length of Stay
Description: Day of life discharged home for untreated and treated infants who completed hospitalization at study site.
  Duration of infant hospitalization-Days
Time Frame: Day of life infants discharged home, which is an expected mean of 21 days.
Population: Untreated and treated infants who completed hospitalization at study site.
Measure: Mean (Standard Deviation); unit: day of life discharged home
Arm/Group | Stochastic Vibrotactile Stimulation (SVS) | Treatment as Usual (TAU)
Number analyzed (Participants) | 94 | 87
day of life discharged home | 11.5 (11.0) | 13.5 (14.6)
Statistical Analysis 1: Comparison: Stochastic Vibrotactile Stimulation (SVS) vs Treatment as Usual (TAU); Test type: Equivalence — A statistical test comparing day of life discharged among untreated infants who completed hospitalization at study site (n=181); p = 0.29, t-test, 2 sided; df = 179 based on number of infants who completed hospitalization at study site

4. Primary Outcome: Hospitalization Length of Stay for Untreated Infants
Description: Day of life discharged home for untreated infants (infants whose Finnegan scores did not meet criteria to treat) who completed hospitalization at study site.
  Duration of infant hospitalization-Days
Time Frame: Day of life untreated infants discharged home, which is an expected mean of 21 days.
Measure: Mean (Standard Deviation); unit: day of life discharged home
Arm/Group | Stochastic Vibrotactile Stimulation (SVS) | Treatment as Usual (TAU)
Number analyzed (Participants) | 65 | 56
day of life discharged home | 5.9 (1.6) | 5.7 (1.3)
Statistical Analysis 1: Comparison: Stochastic Vibrotactile Stimulation (SVS) vs Treatment as Usual (TAU); Test type: Equivalence — A statistical test comparing day of life discharged among untreated infants (n=121); p = 0.55, t-test, 2 sided; df = 119 based on number of infants who did not receive morphine treatment

5. Primary Outcome: Hospitalization Length of Stay for Treated Infants
Description: Day of life discharged home for treated infants (infants whose Finnegan scores met criteria to treat) who completed hospitalization at study site.
  Duration of infant hospitalization-Days
Time Frame: Day of life treated infants discharged home, which is an expected mean of 21 days.
Measure: Mean (Standard Deviation); unit: day of life discharged home
Arm/Group | Stochastic Vibrotactile Stimulation (SVS) | Treatment as Usual (TAU)
Number analyzed (Participants) | 29 | 31
day of life discharged home | 24.1 (12.7) | 27.7 (17.0)
Statistical Analysis 1: Comparison: Stochastic Vibrotactile Stimulation (SVS) vs Treatment as Usual (TAU); Test type: Equivalence — A statistical test comparing day of life discharged among treated infants, n=60; p = 0.36, t-test, 2 sided; df = 58 based on number of infants who received morphine treatment

6. Primary Outcome: Length of Pharmacological Treatment-Duration
Description: For infants who received pharmacotherapy, total days of morphine treatment.
Time Frame: Participants will be monitored for the duration of their hospitalization, which is an expected mean of 21 days
Population: Analyzed cohort who received morphine treatment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Stochastic Vibrotactile Stimulation (SVS) | Treatment as Usual (TAU)
Number analyzed (Participants) | 29 | 31
days | 19.9 (12.7) | 21.6 (9.4)
Statistical Analysis 1: Comparison: Stochastic Vibrotactile Stimulation (SVS) vs Treatment as Usual (TAU); Test type: Equivalence — A test of equivalence was conducted for unadjusted comparisons. A t test of means was used for unadjusted comparisons; p = 0.56, t-test, 2 sided; df = 58 based on number of infants who received morphine treatment

7. Primary Outcome: Trajectory of Symptom Severity Among Treated Infants
Description: Days to start morphine treatment based on Finnegan severity scores among infants who met clinical criteria to treat
Time Frame: Day of life infant started morphine treatment
Measure: Mean (Standard Deviation); unit: day of life started treatment
Arm/Group | Stochastic Vibrotactile Stimulation (SVS) | Treatment as Usual (TAU)
Number analyzed (Participants) | 29 | 31
day of life started treatment | 2.5 (1.2) | 2.9 (1.8)
Statistical Analysis 1: Comparison: Stochastic Vibrotactile Stimulation (SVS) vs Treatment as Usual (TAU); Test type: Equivalence — A statistical test comparing day of life infant started treatment as performed for the cohort that was treated with morphine (n=60); p = 0.25, t-test, 2 sided; df = 58 based on number of infants who received morphine treatment

8. Primary Outcome: Velocity of Weight Gain
Description: Weight loss precedes weight gain in newborns. Days to weight nadir, defined as the lowest weight following birthweight. Velocity of weight gain was measured as days to return to birthweight, i.e., the day on which weight reached or surpassed birthweight following initial weight loss from birth.
Time Frame: Participants will be monitored for the duration of their hospitalization, which is an expected mean of 21 days
Population: Nadir was obtained in treated and untreated infants who completed hospitalization at study site. Weight gain was obtained only in pharmacologically treated infants; untreated infants were discharged prior to weight gain.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Stochastic Vibrotactile Stimulation (SVS) | Treatment as Usual (TAU)
Number analyzed (Participants) | 94 | 87
days
  Nadir | 4.98 (1.49) | 5.05 (1.55)
  Return to Birthweight: number analyzed (Participants) | 24 | 31
  Return to Birthweight | 12.38 (3.87) | 13.48 (4.01)

9. Primary Outcome: Neurobehavioral Outcomes Assessment
Description: Scores for Cognitive Domain Bayley Scales of Infant and Toddler Development Third Edition. The standardized scores have a mean of 100 and standard deviation (SD) of 15. Scores below 1 SD (= or less than 84) is considered below normal. Scores above 1 SD (>115) represent higher than normal functioning.
Time Frame: 6 month and 12 months of life
Population: Study infants who participated in follow-up assessments post hospitalization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stochastic Vibrotactile Stimulation (SVS) | Treatment as Usual (TAU)
Number analyzed (Participants) | 36 | 24
score on a scale
  Cognitive Score at 6 months: number analyzed (Participants) | 28 | 18
  Cognitive Score at 6 months | 99.1 (17.6) | 98.1 (15.6)
  Cognitive Score at 12 months: number analyzed (Participants) | 24 | 17
  Cognitive Score at 12 months | 101.5 (13.1) | 98.8 (13.2)

10. Other Pre Specified Outcome: Respiratory Rate
Description: Respiratory rate at 1 week of age assessed for about 12 consecutive hours in a subset of subjects
Time Frame: Assess respiratory rate for about 12 consecutive hours at week 1 of infant hospitalization
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious and Other adverse events (AE) were obtained for up to 14 months; includes in-hospital and reports obtained post-hospital discharge throughout the follow-up period.
Description: All-Cause Mortality, Serious and Other Adverse events were obtained for both the SVS (intervention) and TAU (control) groups.
  Serious AEs reported include medical events that may occur in NICU environments, e.g. cluster necrotizing enterocolitis (NEC).
  Inherent AEs routinely assessed via Finnegan were not reported; AEs determined by medical caregiver and/or study safety officer that fell outside scope and/or degree of medical events commonly experienced by subject population.
Arm/Group | Stochastic Vibrotactile Stimulation (SVS) | Treatment as Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/105 | 1/103
Serious Adverse Events (participants affected / at risk) | 1/105 | 1/103
Other Adverse Events (participants affected / at risk) | 0/105 | 0/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stochastic Vibrotactile Stimulation (SVS) (N=105) | Treatment as Usual (TAU) (N=103)
cluster necrotizing enterocolitis (Gastrointestinal disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
Enrollment closed at 208 infants before reaching proposed enrollment of 220 infants due to the administration at UMass reneging support for the project, requiring close out at UMass site. PI and funding support were transferred to complete the project at the UPitt site. Delays in reporting reflect transfer-related project restructuring and reduction in study personnel.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/31/NCT02801331/Prot_SAP_000.pdf